CLINICAL TRIAL: NCT04244175
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Trial of CVL-865 as Adjunctive Therapy in Adults With Drug-Resistant Focal Onset Seizures (REALIZE Trial)
Brief Title: A Trial of the Efficacy and Safety of CVL-865 as Adjunctive Therapy in the Treatment of Focal Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-865-SZ-001; 2019-002576-14 (EudraCT Number)
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Seizures
Keywords: CVL-865; Anti-epileptic drugs (AEDs); Focal epilepsy; γ-aminobutyric acid (GABA); Partial seizure; PF-06372865; Darigabat
MeSH Terms: conditions — Seizures; Epilepsies, Partial | interventions — PF-06372865

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received a placebo matched to CVL-865 tablets orally twice a day (BID) during the 2-week Titration Phase, the 8-week Maintenance Phase, and the 3-week Taper Phase.
  Interventions: Drug: Placebo
- CVL-865 7.5 mg BID (Experimental): CVL-865 tablets were administered orally as 2.5 mg twice a day (BID) for 1 week followed by 5 mg BID for another week during the Titration Phase, and then 7.5 mg BID during the 8-week Maintenance Phase. For participants not enrolling into the open-label extension trial, following the Maintenance Phase the dose was gradually decreased over a 3-week Taper Phase.
  Interventions: Drug: CVL-865
- CVL-865 25 mg BID (Experimental): CVL-865 tablets were administered orally as 5 mg twice a day (BID) for 1 week followed by 12.5 mg for another week during the Titration Phase, and then 25 mg BID during the 8-week Maintenance Phase. For participants not enrolling into the open-label extension trial, following the Maintenance Phase the dose was gradually decreased over a 3-week Taper Phase.
  Interventions: Drug: CVL-865

INTERVENTIONS:
Drug: Placebo — Participants received CVL-865 matched placebo tablets orally twice a day (BID) during the Treatment Period.
  Arms: Placebo
Drug: CVL-865 — Participants received CVL-865 tablets orally twice a day (BID) up to the maximum dose of 7.5 mg BID or 25 mg BID during the Treatment Period.
  Other Names: Darigabat; PF-06372865
  Arms: CVL-865 25 mg BID; CVL-865 7.5 mg BID

SUMMARY:
The goal of this clinical trial is to learn if CVL-865, when taken regularly with other anti-seizure medicines, works to prevent seizures in adults with drug-resistant focal onset seizures. It will also learn about the safety of CVL-865.

The main question it aims to answer is whether CVL-865, when taken regularly with other anti-seizure medicines, lowers the number of seizures in those with a diagnosis of epilepsy with drug-resistant focal onset seizures.

This study has an 8-week Screening/Baseline Period, a 13-week Treatment Period (including a 2-week Titration Phase, an 8-week Maintenance Phase, and a 3-week Taper Phase), and a 4-week Safety Follow-Up Period.

Participants will take CVL-865 or a placebo twice a day during the 10-13 week Treatment Period, visit the clinic every few weeks for checkups, tests, and surveys, and fill out an e-Diary.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of epilepsy with focal onset, as defined in the International League Against Epilepsy (ILAE) Classification of Seizures, focal aware (except participants with only focal aware seizures without a motor component), focal impaired awareness, and focal to bilateral tonic-clonic seizures for at least 2 years prior to signing the Informed Consent Form (ICF)
* Participants must have history of an average of 4 or more spontaneous and observable focal onset, as defined in the ILAE Classification of Seizures, focal aware (except participants with only focal aware seizures without a motor component), focal impaired awareness, and focal to bilateral tonic-clonic seizures per 28-day period for at least 3 months (84 days) prior to signing the ICF
* Participants who have tried and failed at least 2 appropriate Anti- epileptic drugs (AEDs) in the past and also currently taking 1 to 3 permitted AEDs at a stable dose for 4 Weeks prior to the Screening Visit
* Participants with a minimum of 8 focal onset, focal aware, focal impaired awareness, or focal to bilateral tonic-clonic seizures during the 8 week baseline period with no 21-day period free of any of these seizure types
* Participants must have had magnetic resonance imaging or contrast enhance computed tomography scan of the brain that demonstrated no progressive structural central nervous system abnormality at the time of the diagnosis of epilepsy
* Participants must have a body mass index (BMI) of 17.5 to 40.0 kilogram per meter square (kg/m^2) and a total body weight greater than (>) 50 kilograms (kg) [110 pounds (lbs)]
* Women of childbearing potential must agree to use an effective method of contraception from signing of informed consent throughout the duration of the study and for 30 days post last dose
* Male must agree to use condom during treatment and until the end of relevant systemic exposure in the male participant for 94 days following the last dose with Investigational Manufacturing Product (IMP)

Exclusion Criteria:

* Participants with (genetic) idiopathic generalized epilepsies or combined generalized and focal epilepsies, including a history of Lennox-Gastaut Syndrome
* Participants with a history of seizures over the past 12 months that occur at such a high frequency they cannot be counted (eg, repetitive seizures, cluster seizures)
* Participants with a history of psychogenic non-epileptic seizures within the year prior to signing the ICF
* Participants with a history of status epilepticus within 5 years prior to signing the ICF
* Participants with a history of neurosurgery for seizures less than 1 year prior to signing the ICF, or radiosurgery less than 2 years prior to signing the ICF
* Participants with a current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological (excluding focal onset epilepsy) disease
* Participants who test positive for human immunodeficiency virus (HIV), hepatitis B and/or or hepatitis C infection
* Participants with a 12-lead ECG demonstrating : QT interval corrected for heart rate using Fridericia's formula >450 milliseconds (msec) (average of 3 ECGs obtained at the Screening Visit); QRS interval >120 msec at the Screening Visit assessed by central reader
* Participants with abnormal laboratory test results which includes (Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) elevated to >2 × Upper limit of normal range (ULN); Total bilirubin greater than or equal to (>=)1.5 × ULN; Females: Hemoglobin <11 gram per deciliter (g/dL); Males: hemoglobin <12 g/dL; White blood cell (WBC) count <3.0 x 10 power 9 per liter (10^9/L); Neutrophil count <2.0 x 10^9/L; Platelet count <150 × 10^9/L
* Use of prohibited medications as listed in the protocol in the absence of appropriate washout phase or the likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Participants taking any drug that is a sensitive P-glycoprotein (P-gp) and Breast cancer resistance protein (BCRP) substrate
* Female participants who are breastfeeding and/or who have a positive pregnancy test result prior to receiving IMP
* Participants who are known to be allergic or hypersensitive to the IMP or any of its components
* Participants who have participated in any clinical trial within 60 days prior to signing the ICF or who have participated in more than 2 clinical trials within the year prior to signing the ICF
* Participants with difficulty swallowing
* Participants who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this CSSRS Item 5 occurred within the last 6 months OR Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred in the last 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (72):
- United States (36):
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Downey, California, Downey, California
  - Loma Linda, California, Loma Linda, California
  - Valencia, California, Valencia, California
  - New Haven, Connecticut, New Haven, Connecticut
  - Altamonte Springs, Florida, Altamonte Springs, Florida
  - Gulf Breeze, Florida, Gulf Breeze, Florida
  - Homestead, Florida, Homestead, Florida
  - Jacksonville, Florida, Jacksonville, Florida
  - Miami, Florida, Miami, Florida
  - Miami Lakes, Florida, Miami Lakes, Florida
  - Orlando, Florida, Orlando, Florida
  - Port Charlotte, Florida, Port Charlotte, Florida
  - Port Orange, Florida, Port Orange, Florida
  - Tampa, Florida, Tampa, Florida
  - Suwanee, Georgia,, Suwanee, Georgia
  - Honolulu, Hawaii, Honolulu, Hawaii
  - Lexington, Kentucky, Lexington, Kentucky
  - Scarborough, Maine, Scarborough, Maine
  - Baltimore, Maryland, Baltimore, Maryland
  - Bethesda, Maryland, Bethesda, Maryland
  - Boston, Massachusetts, Boston, Massachusetts
  - Chesterfield, Missouri, Chesterfield, Missouri
  - Saint Louis, Missouri, St Louis, Missouri
  - Hackensack, New Jersey, Hackensack, New Jersey
  - Mineola, New York, Mineola, New York
  - New York, New York, New York
  - Rochester, New York, Rochester, New York
  - Syracuse, New York, Syracuse, New York
  - Columbus, Ohio, Columbus, Ohio
  - Toledo, Ohio, Toledo, Ohio
  - Oklahoma City, Oklahoma, Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania, Philadelphia, Pennsylvania
  - Charleston, South Carolina, Charleston, South Carolina
  - Nashville, Tennessee, Nashville, Tennessee
  - Salt Lake City, Utah, Salt Lake City, Utah
- Australia (9):
  - Camperdown, New South Wales, Camperdown, New South Wales
  - Randwick, New South Wales, Randwick, New South Wales
  - Westmead, New South Wales, Westmead, New South Wales
  - Herston, Queensland, Herston, Queensland
  - South Brisbane, Queensland, South Brisbane, Queensland
  - Fitzroy, Victoria, Fitzroy, Victoria
  - Heidelberg, Victoria, Heidelberg, Victoria
  - Melbourne, Victoria, Melbourne, Victoria
  - Parkville, Victoria, Parkville, Victoria
- Poland (9):
  - Bydgoszcz, Kujawsko-Pomorskie, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Kraków, Malopolskie, Krakow, Lesser Poland Voivodeship
  - Warszawa, Mazowieckie, Warsaw, Masovian Voivodeship
  - Gdańsk, Pomorskie, Gdansk, Pomeranian Voivodeship
  - Wojnicz, Lskie, Wojnicz, Wojnicz Lskie
  - Białystok, Bialystok
  - Lublin, Lublin
  - Warszawa, Warsaw
  - Lodz, Lodz, Łódź Voivodeship
- Serbia (5):
  - Kragujevac, Sumadija, Kragujevac, Sumadija
  - Neurology Department, Kragujevac, Kragujevac, Sumadija
  - Belgrade, Belgrade
  - Clinic of Neurology, Belgrade, Belgrade
  - Niš, Niš
- South Korea (2):
  - Gwangjin-gu, Seoul, Gwangju, Seoul
  - Irwon-Ro Gangnam-gu., Seoul, Irwon-dong, Seoul
- Spain (8):
  - Malaga,, Málaga, Andalusia
  - Barcelona, Catalunya, Barcelona, Catalonia
  - Terrassa, Terrassa, Catalonia
  - Navarra, Navarro, Navarre
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Sevilla, Seville
  - Valencia, Valencia
- Ukraine (3):
  - Uzhgorod, Uzhhorod, Uzhgorod
  - Kyiv, Kyiv
  - Lviv, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurrell R, Iredale P, Evrard A, Duveau V, Ruggiero C, Roucard C. Pronounced antiseizure activity of the subtype-selective GABAA positive allosteric modulator darigabat in a mouse model of drug-resistant focal epilepsy. CNS Neurosci Ther. 2022 Nov;28(11):1875-1882. doi: 10.1111/cns.13927. Epub 2022 Aug 14. PMID 35965432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 62 sites in 7 countries.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to one of three treatment groups: Placebo, CVL-865 7.5 mg twice a day (BID), and CVL-865 25 mg BID.
Period: Overall Study
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID
Started | 51 | 51 | 52
Completed | 44 | 44 | 42
Not Completed | 7 | 7 | 10
Not completed — Adverse Event | 3 | 2 | 5
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 1
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Other, not specified | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | Total
Number analyzed (Participants) | 51 | 51 | 52 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13.38) | 41.4 (11.04) | 43.1 (12.88) | 41.6 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 23 | 80
  Male | 22 | 23 | 29 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 9 | 21
  Not Hispanic or Latino | 46 | 43 | 42 | 131
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 3 | 5
  Black or African American | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 2 | 5
  White | 46 | 46 | 42 | 134
  Other | 1 | 2 | 1 | 4
  Multiple | 0 | 0 | 1 | 1
Duration of Epilepsy [Mean (Standard Deviation); unit: years] — Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
  years
    number analyzed (Participants) | 51 | 50 | 52 | 153
    (all) | 25.88 (14.595) | 22.98 (14.896) | 23.54 (13.335) | 24.14 (14.243)

OUTCOME MEASURES:

1. Primary Outcome: Response Ratio (RRatio)
Description: Response Ratio (RRatio) is calculated as RRatio=(T-B)/(T+B) ×100, where T represents the focal onset seizure frequency rate per week in the Maintenance Phase and B represents the focal onset seizure frequency rate per week in the Baseline Period. The Response Ratio ranges between -100 and 100; negative values indicate reduction in seizure rate and positive values indicate increase in seizure rate during treatment.
Time Frame: Baseline Period; Maintenance Phase Days 15 through 71
Population: Modified intent-to-treat (mITT): All randomized participants who receive at least 1 dose of investigational medicinal product and have both Baseline seizure frequency recorded in the eDiary with entry compliance ≥20% and at least 1 post-Baseline entry in the seizure diary during the Maintenance Phase. Data are presented for participants with a non-missing value.
Measure: Mean (Standard Deviation); unit: RRatio
Groups:
- CVL-865 7.5 mg BID / 25 mg BID: 7.5 mg BID: CVL-865 tablets were administered orally as 2.5 mg twice a day (BID) for 1 week followed by 5 mg BID for another week during the Titration Phase, and then 7.5 mg BID during the 8-week Maintenance Phase.
  25 mg BID: CVL-865 tablets were administered orally as 5 mg twice a day (BID) for 1 week followed by 12.5 mg for another week during the Titration Phase, and then 25 mg BID during the 8-week Maintenance Phase.
  For participants not enrolling into the open-label extension trial, following the Maintenance Phase the dose was gradually decreased over a 3-week Taper Phase.
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
RRatio | -24.06 (33.441) | -22.45 (26.393) | -25.90 (33.428) | -24.19 (30.041)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo; Test type: Superiority — RRatio was analyzed using an analysis of covariance (ANCOVA) model including treatment and the Baseline seizure frequency per week as a covariate; p = 0.986, ANCOVA; LS Mean Difference = 0.11, 90% CI 2-sided [-10.38 to 10.61] — CVL-865 25 mg BID - Placebo
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.823, ANCOVA; LS Mean Difference = 1.42, 90% CI 2-sided [-9.04 to 11.87] — CVL-865 7.5 mg BID - Placebo
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.888, ANCOVA; LS Mean Difference = 0.76, 90% CI 2-sided [-8.23 to 9.76] — CVL-865 7.5 mg BID / 25 mg BID - Placebo

2. Secondary Outcome: Percentage Change From Baseline in Focal Onset Seizure Frequency Per Week Over the Maintenance Phase
Description: Seizure frequency is defined as the total number of focal onset seizures over the treatment period of interest divided by the total number of days with no missing seizure counts in the corresponding period multiplied by 7.
Time Frame: Baseline Period; Maintenance Phase Days 15 through 71
Population: Modified intent-to-treat (mITT): All randomized participants who receive at least 1 dose of investigational medicinal product and have both Baseline seizure frequency recorded in the eDiary with entry compliance ≥20% and at least 1 post-Baseline entry in the seizure diary during the Maintenance Phase. Data are presented for participants with a non-missing value. Data are presented for participants with a non-missing value.
Measure: Number; unit: Percentage change from Baseline
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
Percentage change from Baseline | -26.2 | -27.2 | -29.8 | -28.5
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo; Test type: Superiority — The percent reduction relative to Placebo was calculated; Percent reduction relative to Placebo = 4.9, 90% CI 2-sided [-12.0 to 19.3]
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo; Test type: Superiority — The percent reduction relative to Placebo was calculated; Percent reduction relative to Placebo = 1.4, 90% CI 2-sided [-16.1 to 16.2]
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo; Test type: Superiority — The percent reduction relative to Placebo was calculated; Percent reduction relative to Placebo = 3.2, 90% CI 2-sided [-11.4 to 15.8]

3. Secondary Outcome: Percentage of Participants With 50 Percent (%) Responder Rate
Description: The 50% responder rate is defined as the percentage of participants with at least a 50% reduction in focal onset seizure frequency rate in the Maintenance Phase compared to the Baseline Period.
Time Frame: Baseline Period; Maintenance Phase Days 15 through 71
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
percentage of participants | 30.0 | 34.8 | 38.3 | 36.6
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo; Test type: Superiority — A logistic regression with treatment group and Baseline seizure frequency as covariates was used to calculate the Odds ratio, 90% confidence interval, and p-value; p = 0.587, Regression, Logistic; Odds Ratio (OR) = 1.270, 90% CI 2-sided [0.616 to 2.618]
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.554, Regression, Logistic; Odds Ratio (OR) = 1.303, 90% CI 2-sided [0.624 to 2.723]
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.513, Regression, Logistic; Odds Ratio (OR) = 1.286, 90% CI 2-sided [0.684 to 2.420]

4. Secondary Outcome: Percentage of Seizure-free Participants During the Maintenance Phase
Description: Seizure freedom is defined as no seizures during the Maintenance Phase.
Time Frame: Maintenance Phase Days 15 through 71
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
percentage of participants | 6.0 | 2.2 | 4.3 | 3.2
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo; Test type: Superiority — The p-value is from Fisher's exact test for number of responders; p > 0.999, Fisher's exact test
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo; Test type: Superiority — The p-value is from Fisher's exact test for number of responders; p = 0.618, Fisher's exact test
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo; Test type: Superiority — The p-value is from Fisher's exact test for number of responders; p = 0.422, Fisher's exact test

5. Secondary Outcome: Weekly Seizure Rate During the Maintenance Phase
Description: as for outcome 2
Time Frame: Maintenance Phase Weeks 1, 2, 3, 4, 5, 6, 7, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seizures/week
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
Seizures/week
  Maintenance Phase Week 1 | 6.41 (10.772) | 5.20 (5.867) | 2.71 (4.804) | 3.95 (5.472)
  Maintenance Phase Week 2: number analyzed (Participants) | 48 | 45 | 47 | 92
  Maintenance Phase Week 2 | 5.66 (8.858) | 4.98 (5.982) | 2.74 (4.506) | 3.84 (5.370)
  Maintenance Phase Week 3: number analyzed (Participants) | 49 | 45 | 46 | 91
  Maintenance Phase Week 3 | 6.81 (10.391) | 6.53 (9.010) | 3.26 (5.018) | 4.88 (7.414)
  Maintenance Phase Week 4: number analyzed (Participants) | 47 | 45 | 45 | 90
  Maintenance Phase Week 4 | 6.20 (8.888) | 6.44 (9.974) | 3.29 (5.130) | 4.87 (8.044)
  Maintenance Phase Week 5: number analyzed (Participants) | 45 | 45 | 44 | 89
  Maintenance Phase Week 5 | 5.76 (9.269) | 6.27 (8.688) | 3.21 (6.111) | 4.75 (7.639)
  Maintenance Phase Week 6: number analyzed (Participants) | 45 | 45 | 43 | 88
  Maintenance Phase Week 6 | 5.44 (9.939) | 6.21 (8.313) | 3.29 (6.070) | 4.79 (7.408)
  Maintenance Phase Week 7: number analyzed (Participants) | 45 | 45 | 42 | 87
  Maintenance Phase Week 7 | 5.96 (9.864) | 6.40 (8.520) | 4.65 (8.235) | 5.56 (8.381)
  Maintenance Phase Week 8: number analyzed (Participants) | 42 | 44 | 40 | 84
  Maintenance Phase Week 8 | 6.62 (10.797) | 5.23 (6.883) | 3.60 (7.063) | 4.45 (6.975)

6. Secondary Outcome: Patient's Global Impression of Change (PGI-C) Score at Maintenance Phase Days 15, 43, and 71
Description: The self-report measure Patient's Global Impression of Change (PGI-C) reflects a participant's belief about the efficacy of treatment. It is a 7-point scale depicting a participant's rating of overall improvement where 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse and 7 = very much worse. Lower scores indicate improvement.
Time Frame: Maintenance Phase Days 15, 43, and 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
units on a scale
  Maintenance Phase Day 15 | 3.5 (0.76) | 3.3 (0.96) | 3.0 (1.27) | 3.1 (1.13)
  Maintenance Phase Day 43: number analyzed (Participants) | 48 | 46 | 47 | 93
  Maintenance Phase Day 43 | 3.5 (1.11) | 3.2 (1.06) | 3.0 (1.41) | 3.1 (1.24)
  Maintenance Phase Day 71: number analyzed (Participants) | 45 | 45 | 42 | 87
  Maintenance Phase Day 71 | 3.3 (1.00) | 3.0 (1.02) | 3.0 (1.36) | 3.0 (1.19)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 15); Test type: Superiority — The PGI-C score over time was analyzed using a Mixed Model for Repeated Measures (MMRM) analysis. Treatment group, visit, and the interaction between treatment group and visit was included as fixed factors in the MMRM. Participant was included as a random effect, and an unstructured covariance structure was used for the repeated measures; p = 0.021, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.5, 90% CI 2-sided [-0.8 to -0.1] — CVL-865 25 mg BID - Placebo (Day 15)
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.342, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.2, 90% CI 2-sided [-0.5 to 0.1] — CVL-865 7.5 mg BID - Placebo (Day 15)
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.059, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.6 to 0.0] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 15)
Statistical Analysis 4: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.040, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.5, 90% CI 2-sided [-0.9 to -0.1] — CVL-865 25 mg BID - Placebo (Day 43)
Statistical Analysis 5: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.152, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 90% CI 2-sided [-0.8 to 0.1] — CVL-865 7.5 mg BID - Placebo (Day 43)
Statistical Analysis 6: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.044, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 90% CI 2-sided [-0.8 to -0.1] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 43)
Statistical Analysis 7: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.199, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.7 to 0.1] — CVL-865 25 mg BID - Placebo (Day 71)
Statistical Analysis 8: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.171, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.7 to 0.1] — CVL-865 7.5 mg BID - Placebo (Day 71)
Statistical Analysis 9: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.125, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.7 to 0.0] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 71)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Symptoms Scale (CGI-S) Score at Maintenance Phase Days 15, 43, and 71
Description: The CGI-S is an observer-rated scale that was used to measure symptom severity. It is a 7-point scale depicting a participants rating of overall improvement. Participants rate their change as 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Maintenance Phase Days 15, 43, and 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 45 | 91
units on a scale
  Maintenance Phase Day 15 | -0.2 (0.66) | 0.0 (0.94) | -0.3 (0.87) | -0.2 (0.92)
  Maintenance Phase Day 43: number analyzed (Participants) | 49 | 46 | 45 | 91
  Maintenance Phase Day 43 | -0.2 (0.97) | -0.2 (1.05) | -0.6 (0.91) | -0.4 (1.00)
  Maintenance Phase Day 71: number analyzed (Participants) | 44 | 45 | 39 | 84
  Maintenance Phase Day 71 | -0.3 (0.97) | -0.3 (1.09) | -0.7 (1.09) | -0.5 (1.10)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 15); Test type: Superiority — The CGI-S score over time was analyzed using a Mixed Model for Repeated Measures (MMRM) analysis. Treatment group, visit, and the interaction between treatment group and visit was included as fixed factors in the MMRM. Participant was included as a random effect, and an unstructured covariance structure was used for the repeated measures; p = 0.767, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.2] — CVL-865 25 mg BID - Placebo (Day 15)
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.178, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.2, 90% CI 2-sided [0.0 to 0.5] — CVL-865 7.5 mg BID - Placebo (Day 15)
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.542, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 90% CI 2-sided [-0.1 to 0.3] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 15)
Statistical Analysis 4: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.106, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.6 to 0.0] — CVL-865 25 mg BID - Placebo (Day 43)
Statistical Analysis 5: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.663, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.1, 90% CI 2-sided [-0.2 to 0.4] — CVL-865 7.5 mg BID - Placebo (Day 43)
Statistical Analysis 6: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.488, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.2] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 43)
Statistical Analysis 7: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.100, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.7 to 0.0] — CVL-865 25 mg BID - Placebo (Day 71)
Statistical Analysis 8: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.969, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = 0.0, 90% CI 2-sided [-0.3 to 0.3] — CVL-865 7.5 mg BID - Placebo (Day 71)
Statistical Analysis 9: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.344, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.2, 90% CI 2-sided [-0.4 to 0.1] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 71)

8. Secondary Outcome: Clinical Global Impression-Improvement Scale (CGI-I) Score at Maintenance Phase Days 15, 43, and 71
Description: The CGI-I is an observer-rated scale that was used to measure the participant's symptom severity compared with before initiation of treatment with the investigational medicinal product (IMP). It is a 7-point scale depicting a participant's change from Baseline in symptom severity using the following response choices: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Lower scores indicate improvement.
Time Frame: Baseline, Maintenance Phase Days 15, 43, and 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 50 | 46 | 47 | 93
units on a scale
  Maintenance Phase Day 15 | 3.5 (0.71) | 3.4 (0.83) | 3.1 (0.91) | 3.2 (0.88)
  Maintenance Phase Day 43: number analyzed (Participants) | 49 | 46 | 47 | 93
  Maintenance Phase Day 43 | 3.5 (0.84) | 3.3 (1.02) | 2.9 (1.23) | 3.1 (1.15)
  Maintenance Phase Day 71: number analyzed (Participants) | 45 | 43 | 41 | 84
  Maintenance Phase Day 71 | 3.3 (0.96) | 3.3 (0.98) | 2.8 (1.46) | 3.0 (1.25)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 15); Test type: Superiority — The CGI-I score over time was analyzed using a Mixed Model for Repeated Measures (MMRM) analysis. Treatment group, visit, and the interaction between treatment group and visit was included as fixed factors in the MMRM. Participant was included as a random effect, and an unstructured covariance structure was used for the repeated measures; p = 0.010, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 90% CI 2-sided [-0.7 to -0.2] — CVL-865 25 mg BID - Placebo (Day 15)
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.376, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 90% CI 2-sided [-0.4 to 0.1] — CVL-865 7.5 mg BID - Placebo (Day 15)
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 15); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.044, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.3, 90% CI 2-sided [-0.5 to -0.1] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 15)
Statistical Analysis 4: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.005, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.6, 90% CI 2-sided [-1.0 to -0.3] — CVL-865 25 mg BID - Placebo (Day 43)
Statistical Analysis 5: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.549, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.2] — CVL-865 7.5 mg BID - Placebo (Day 43)
Statistical Analysis 6: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 43); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.048, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 90% CI 2-sided [-0.7 to -0.1] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 43)
Statistical Analysis 7: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.005, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.6, 90% CI 2-sided [-1.0 to -0.3] — CVL-865 25 mg BID - Placebo (Day 71)
Statistical Analysis 8: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.549, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.1, 90% CI 2-sided [-0.5 to 0.2] — CVL-865 7.5 mg BID - Placebo (Day 71)
Statistical Analysis 9: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (Day 71); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.048, Mixed Model for Repeated Measures (MMRM); LS Mean Difference = -0.4, 90% CI 2-sided [-0.7 to -0.1] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (Day 71)

9. Secondary Outcome: Change From Baseline in Quality of Life in Epilepsy-31 (QOLIE-31) Overall Score at Maintenance Phase Day 71
Description: The Quality of Life in Epilepsy-31 (QOLIE-31) contains 7 multi-item scales that cover the following health concepts: emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, and overall quality of life. A QOLIE-31 overall score is obtained using a weighted average of the multi-item scale scores. The QOLIE-31 also includes a single item that assessed overall health. The QOLIE-31 score range is from 0 to 100 with a higher score indicating a better outcome for quality of life. Positive changes from Baseline indicate improvement.
Time Frame: Baseline, Maintenance Phase Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 46 | 44 | 46 | 90
units on a scale | 0.29 (9.859) | 2.08 (12.717) | 3.70 (12.267) | 2.91 (12.445)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo; Test type: Superiority — Changes from Baseline in QOLIE-31 Overall Scores was compared using an ANCOVA model with the Baseline score as a covariate and treatment group included in the model as fixed effects in the mITT population. This estimand included available post-Baseline response data that occurred before discontinuation of treatment or the addition of rescue medication; p = 0.829, ANCOVA; LS Mean Difference = -0.49, 90% CI 2-sided [-4.23 to 3.26] — CVL-865 25 mg BID - Placebo
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.927, ANCOVA; LS Mean Difference = -0.20, 90% CI 2-sided [-3.87 to 3.46] — CVL-865 7.5 mg BID - Placebo
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.859, ANCOVA; LS Mean Difference = -0.35, 90% CI 2-sided [-3.57 to 2.88] — CVL-865 7.5 mg BID / 25 mg BID - Placebo

10. Secondary Outcome: Change From Baseline in Health Utilities Index (HUI) Utility Score at Maintenance Phase Day 71
Description: The Health Utilities Index (HUI) is a rating scale used to measure general health status and health-related quality of life. In HUI, utility values range from -0.03 and -0.36 for the HUI-2 and HUI-3, respectively, to 1.00. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Maintenance Phase Day 71
Population: Modified intent-to-treat (mITT): All randomized participants who receive at least 1 dose of investigational medicinal product and have both Baseline seizure frequency recorded in the eDiary with entry compliance ≥20% and at least 1 post Baseline entry in the seizure diary during the Maintenance Phase. Data are presented for participants with a non-missing value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 48 | 44 | 46 | 90
units on a scale
  HUI-2 | -0.029 (0.2579) | 0.052 (0.2162) | -0.014 (0.3084) | 0.018 (0.2679)
  HUI-3 | -0.025 (0.3961) | 0.110 (0.3448) | -0.012 (0.4469) | 0.048 (0.4027)
Statistical Analysis 1: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (HUI-2); Test type: Superiority — The Least Square Means (LS Means), difference in LS Means, 90% confidence interval for the difference, and the p-value for the difference are from an analysis of covariance (ANCOVA) model with fixed effects for treatment and Baseline score; p = 0.788, ANCOVA; LS Mean Difference = -0.013, 90% CI 2-sided [-0.096 to 0.069] — CVL-865 25 mg BID - Placebo (HUI-2)
Statistical Analysis 2: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (HUI-2); Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.126, ANCOVA; LS Mean Difference = 0.077, 90% CI 2-sided [-0.006 to 0.160] — CVL-865 7.5 mg BID - Placebo (HUI-2)
Statistical Analysis 3: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (HUI-2); Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.461, ANCOVA; LS Mean Difference = 0.032, 90% CI 2-sided [-0.039 to 0.103] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (HUI-2)
Statistical Analysis 4: Comparison: Placebo vs CVL-865 25 mg BID; CVL-865 25 mg BID vs Placebo (HUI-3); Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.661, ANCOVA; LS Mean Difference = -0.032, 90% CI 2-sided [-0.154 to 0.089] — CVL-865 25 mg BID - Placebo (HUI-3)
Statistical Analysis 5: Comparison: Placebo vs CVL-865 7.5 mg BID; CVL-865 7.5 mg BID vs Placebo (HUI-3); Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.124, ANCOVA; LS Mean Difference = 0.115, 90% CI 2-sided [-0.008 to 0.237] — CVL-865 7.5 mg BID - Placebo (HUI-3)
Statistical Analysis 6: Comparison: Placebo vs CVL-865 7.5 mg BID / 25 mg BID; CVL-865 7.5 mg BID / 25 mg BID vs Placebo (HUI-3); Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.518, ANCOVA; LS Mean Difference = 0.041, 90% CI 2-sided [-0.064 to 0.146] — CVL-865 7.5 mg BID / 25 mg BID - Placebo (HUI-3)

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Any TEAE | 28 | 33 | 46 | 79
  TESAE | 1 | 4 | 1 | 5

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECGs)
Description: 12-lead electrocardiogram (ECG) recordings were obtained after the participant had been supine and at rest for at least 5 minutes.
Time Frame: Baseline; From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Absolute QTcF Interval (msec), > 450 and ≤480 msec | 0 | 1 | 2 | 3
  Absolute QTcF Interval (msec), > 480 and ≤500 msec | 0 | 0 | 0 | 0
  Absolute QTcF Interval (msec), > 500 msec | 0 | 0 | 0 | 0
  Change from Baseline in QTcF Interval, > 30 - 60 msec | 4 | 2 | 1 | 3
  Change from Baseline in QTcF Interval, > 60 msec | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: Vital signs were measured with the participant in a sitting/semi-recumbent position after 5 minutes rest and included temperature, systolic and diastolic blood pressure, respiratory rate, and heart rate.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Systolic Blood Pressure < 90 mmHg | 0 | 1 | 0 | 1
  Systolic Blood Pressure > 140 mmHg | 4 | 0 | 1 | 1
  Diastolic Blood Pressure < 50 mmHg | 0 | 1 | 0 | 1
  Diastolic Blood Pressure > 90 mmHg | 4 | 0 | 2 | 2
  Heart Rate < 60 beats/min | 6 | 6 | 14 | 20
  Heart Rate > 100 beats/min | 2 | 1 | 0 | 1
  Respiratory Rate < 12 breaths/min | 0 | 0 | 0 | 0
  Respiratory Rate > 20 breaths/min | 0 | 0 | 1 | 1
  Temperature < 36 °C | 2 | 2 | 7 | 9
  Temperature > 38 °C | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results
Description: The number of participants with clinically significant changes in physical and neurological examination results was documented.
Time Frame: Baseline; From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Clinically Significant Changes in Physical Examination | 3 | 1 | 2 | 3
  Clinically Significant Changes in Neurological Examination | 5 | 1 | 5 | 6

15. Secondary Outcome: Number of Participants With Positive Response to Columbia Suicide-Severity Rating Scale (C-SSRS)
Description: The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Suicidal Ideation: (1) Wish to be dead | 0 | 0 | 2 | 2
  Suicidal Ideation: (2) Non-specific active suicidal thoughts | 0 | 0 | 1 | 1
  Suicidal Ideation: (3) Active suicidal ideation with any methods (not plan) without intent to act | 0 | 1 | 0 | 1
  Suicidal Ideation: (4) Active suicidal ideation with some intent to act, without specific plan | 0 | 0 | 0 | 0
  Suicidal Ideation: (5) Active suicidal ideation with specific plan and intent | 0 | 0 | 0 | 0

16. Secondary Outcome: Change in Modified Clinical Institute Withdrawal Assessment - Benzodiazepines (mCIWA-B) From Last On-treatment Assessment
Description: The modified Clinical Institute Withdrawal Assessment - Benzodiazepines (mCIWA-B) is a sensitive instrument to measure withdrawal under conditions where there is a taper of medication (rather than abrupt discontinuation). It consists of 17-items that monitor the type and severity of BZD withdrawal symptoms such as irritability, fatigue, appetite, and sleeplessness. The total score ranges from 1 to 68 with higher scores indicating more severe withdrawal. Baseline is defined as the last on-treatment assessment on Day 71. Negative changes from Baseline indicate a reduction in withdrawal symptoms.
Time Frame: Maintenance Phase Day 71, Taper Phase Days 78, 85, and 92, and Safety Follow-up Days 99 and 120
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP). Data are presented for participants with a non-missing value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 7 | 10 | 10 | 20
units on a scale
  Taper Phase Day 78 | -0.9 (3.13) | 0.7 (3.09) | -1.0 (1.87) | -0.1 (2.66)
  Taper Phase Day 85 | -1.7 (3.35) | -0.4 (5.64) | -0.2 (3.56) | -0.3 (4.64)
  Taper Phase Day 92 | -1.1 (4.85) | -0.5 (4.20) | 1.1 (3.66) | 0.3 (3.93)
  Safety Follow-up Day 99 | -1.7 (5.31) | -0.8 (6.65) | 2.3 (5.79) | 0.7 (6.29)
  Safety Follow-up Day 120 | -1.0 (5.10) | -0.2 (6.09) | 0.9 (4.31) | 0.4 (5.16)

17. Secondary Outcome: Number of Participants With Adverse Events That Are Abuse-related or Involve Medication Handling Irregularities (MHI)
Description: Adverse events potentially related to abuse or dependence of the investigational medicinal product (IMP) were documented.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to Day 120)
Population: Full analysis set: All randomized participants who receive at least 1 dose of investigational medicinal product (IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID | CVL-865 7.5 mg BID / 25 mg BID
Number analyzed (Participants) | 51 | 50 | 52 | 102
Participants
  Abuse-related AEs | 9 | 10 | 20 | 30
  AEs related to Medication Handling Irregularities | 0 | 0 | 0 | 0

18. Secondary Outcome: Plasma Concentrations of CVL-865 on Maintenance Phase Days 15, 43, and 71, and Taper Phase Day 92
Description: Plasma concentration of CVL-865 was measured on Maintenance Phase Days 15, 43, and 71, and Taper Phase Day 92.
Time Frame: Maintenance Phase Days 15, 43, and 71, and Taper Phase Day 92
Population: All randomized participants who receive at least 1 dose of the investigational medicinal product (IMP) and have at least 1 measurable CVL-865 concentration. Data are presented for participants with a non-missing value.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CVL-865 7.5 mg BID | CVL-865 25 mg BID
Number analyzed (Participants) | 44 | 48
ng/mL
  Maintenance Phase Day 15: number analyzed (Participants) | 43 | 48
  Maintenance Phase Day 15 | 30.99 (29.086) | 69.64 (56.166)
  Maintenance Phase Day 43: number analyzed (Participants) | 42 | 46
  Maintenance Phase Day 43 | 34.60 (33.554) | 151.63 (125.931)
  Maintenance Phase Day 71: number analyzed (Participants) | 44 | 41
  Maintenance Phase Day 71 | 32.45 (29.433) | 167.96 (160.999)
  Taper Phase Day 92: number analyzed (Participants) | 11 | 10
  Taper Phase Day 92 | 9.74 (14.978) | 29.02 (34.133)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time informed consent was signed to the end of the study. The median time on follow-up was 127 days for the Placebo group,129 days for the CVL-865 7.5 mg BID group, and 127 days for the CVL-865 25 mg BID group.
Arm/Group | Placebo | CVL-865 7.5 mg BID | CVL-865 25 mg BID
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/51 | 4/51 | 2/52
Other Adverse Events (participants affected / at risk) | 24/51 | 26/51 | 38/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | CVL-865 7.5 mg BID (N=51) | CVL-865 25 mg BID (N=52)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCLONUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | CVL-865 7.5 mg BID (N=51) | CVL-865 25 mg BID (N=52)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 5 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 4 (4)
VISION BLURRED (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 2 (3)
FATIGUE (General disorders) | 2 (2) | 3 (6) | 6 (6)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 5 (8) | 3 (3) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (3)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
DIZZINESS (Nervous system disorders) | 4 (4) | 3 (4) | 10 (10)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 3 (3) | 4 (8) | 6 (12)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 4 (4) | 6 (7) | 7 (7)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4)
APATHY (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 5 (5) | 1 (1) | 2 (2)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT04244175/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT04244175/SAP_001.pdf